CLINICAL TRIAL: NCT04464460
Title: A Randomized, Double-blind, Placebo-Controlled Multicenter Phase 1b Study to Evaluate the Safety, Pharmacokinetics, and Efficacy of 2 Different Intravenous Doses of TAK-671 for the Treatment of Coronavirus Disease 2019 in Adults
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics (PK), and Efficacy of TAK-671 for the Treatment of Coronavirus Disease (COVID) 2019 in Adults
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Decision (no enrollment)
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-671-1501; U1111-1252-9426 (Registry Identifier: WHO)
Record Dates: First submitted 2020-07-08; First posted 2020-07-09 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Coronavirus Disease
Keywords: Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: TAK-671 Low Dose (Experimental): TAK-671 low dose or TAK-671 placebo-matching, infusion over a 90-minute period, intravenously, once on Day 1.
  Interventions: Drug: TAK-671; Drug: TAK-671 Placebo
- Cohort 2: TAK-671 High Dose (Experimental): TAK-671 high dose or TAK-671 placebo-matching, infusion over a 90-minute period, intravenously, once on Day 1.
  Interventions: Drug: TAK-671; Drug: TAK-671 Placebo

INTERVENTIONS:
Drug: TAK-671 — TAK-671 intravenous infusion.
  Other Names: SB26
Drug: TAK-671 Placebo — TAK-671 placebo-matching intravenous infusion.
  Other Names: SB26/TAK-671 matching-placebo

SUMMARY:
The purpose of this study is to assess safety, tolerability, preliminary efficacy, and PK of TAK-671 in participants with COVID-19.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-671. The study will evaluate the safety, tolerability and PK of TAK-671 in participants admitted to the hospital with a confirmed severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) positive test.

The study will enroll approximately 40 participants. Each cohort will have 20 participants. Participants will be randomly assigned (by chance, like flipping a coin) in a 3:1 ratio to receive TAK-671 or placebo in each cohort, which will remain undisclosed to the participant during the study (unless there is an urgent medical need):

* Cohort 1: TAK-671 Low Dose
* Cohort 2: TAK-671 High Dose

Enrollment in Cohort 2 will only begin once all 20 participants in Cohort 1 have reached Day 7 post dose and have received positive review from the internal review committee (IRC) and approval to continue enrollment. All participants will receive the standard of care along with the study treatment.

This multi-center trial will be conducted in the United States. The overall time to participate in this study is approximately 3 months. All participants will be followed up 28 days after the infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Has laboratory-confirmed SARS-CoV-2 infection as determined via polymerase chain reaction or an accepted molecular assay of any specimen, example, respiratory, blood, urine, stool, other body fluid.
2. It has been less than 72 hours since time of the participant's hospital admission, or, if hospital acquired COVID-19 is confirmed, less than 72 hours after confirmation of positive SARS-CoV-2 test or the onset of respiratory symptoms, whichever is first.
3. Has peripheral capillary SpO2 less than or equal to 93% on room air.
4. Weighs greater than or equal to (>=) 50 kilogram (kg) and has a body mass index (BMI) 18 to 35 kilogram per square meter (kg/m^2), inclusive.
5. Female participants are post-menopausal or surgically sterile.

Exclusion Criteria:

1. Has received TAK-671 or ulinastatin (UTI) in a previous clinical study or as a therapeutic agent.
2. Has received a human blood product (other than a transfusion needed for trauma treatment) or has been treated with a monoclonal antibody or Fc-fusion biologic within 5 years of the screening visit.
3. Has evidence of multiorgan failure, based on a SOFA score greater than 12.
4. Is on invasive mechanical ventilation.
5. Requires vasopressor support. (However, use of fluid support is not exclusionary.)
6. Has known or suspected venous thromboembolism.
7. Any female participant who is of child-bearing potential or is breastfeeding.
8. Has active tuberculosis or a clinical suspicion of latent tuberculosis.
9. Has fulminant hepatic or renal failure.
10. Has congestive heart failure of New York Heart Association Grade III or IV, pulmonary embolism, or any other serious cardiac condition (example, pericardial effusion or restrictive cardiomyopathy).
11. Participant's progression to death is imminent and inevitable within the next 24 hours, regardless of cause and irrespective of the provision of treatments, in the opinion of the investigator.
12. Has a life expectancy of less than 6 months due to reasons other than COVID-19 in the opinion of the investigator.
13. Has a do-not-resuscitate or do-not-intubate (DNR/DNI) order.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-25 (Estimated); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs) | Baseline up to Day 28
Number of Participants With Markedly Abnormal Laboratory Values | Baseline up to Day 28
Number of Participants With Markedly Abnormal Values of Vital Signs | Baseline up to Day 28
Number of Participants With Markedly Abnormal 12-lead Electrocardiograms | Baseline up to Day 28
Number of Participants With Adverse Events (AEs) Related to Physical Examination Findings | Baseline up to Day 28
Ceoi: Serum Concentration at the end of Infusion for TAK-671 | Day 14: at the end of infusion (at 336 hours post infusion)
T1/2z: Terminal Disposition Serum Half-life for TAK-671 | Day 0 pre-infusion and at multiple time points (up to 336 hours) post-infusion
AUClast: Area Under the Serum Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-671 | Day 0 pre-infusion and at multiple time points (up to 336 hours) post-infusion
AUC∞: Area Under the Serum Concentration-time Curve From Time 0 to Infinity for TAK-671 | Day 0 pre-infusion and at multiple time points (up to 336 hours) post-infusion

SECONDARY OUTCOMES:
Percentage of Participants With Sustained Clinical Improvement or Live Discharge at Day 28 | Day 28
  Sustained clinical improvement is defined as a 2-point improvement on the 8-point ordinal scale for clinical improvement, that is at least 2 points increase from the lowest score recorded since randomization and no worsening of the score afterwards by Day 28. An 8-point ordinal scale for clinical improvement in COVID-19 symptoms ranges from a score of 1 to a score of 8, where 1 (death), 2 (hospitalized, on invasive mechanical ventilation or ECMO), 3 (hospitalized, on non-invasive ventilation or high-flow oxygen devices), 4 (hospitalized, requiring supplemental oxygen), 5 (hospitalized, not requiring supplemental oxygen, requiring ongoing medical care [COVID-19 related or otherwise]), 6 (hospitalized, not requiring supplemental oxygen, no longer requires ongoing medical care), 7 (not hospitalized, limitation on activities and/or requiring home oxygen), and 8 (not hospitalized, no limitations on activities).
Percentage of Participants With Sustained Clinical Recovery | Up to 28 days
  Sustained clinical recovery is defined as achieving score 6, 7, or 8 based on the ordinal scale and maintained the clinical recovery until Day 28. An 8-point ordinal scale for clinical improvement in COVID-19 symptoms ranges from a score of 1 to a score of 8, where 1 (death), 2 (hospitalized, on invasive mechanical ventilation or ECMO), 3 (hospitalized, on non-invasive ventilation or high-flow oxygen devices), 4 (hospitalized, requiring supplemental oxygen), 5 (hospitalized, not requiring supplemental oxygen, requiring ongoing medical care [COVID-19 related or otherwise]), 6 (hospitalized, not requiring supplemental oxygen, no longer requires ongoing medical care), 7 (not hospitalized, limitation on activities and/or requiring home oxygen), and 8 (not hospitalized, no limitations on activities).
Percentage of Participants With Sustained Remission of Respiratory Symptoms | Up to 28 days
  Sustained remission of respiratory symptoms is defined as independence from supplemental oxygen therapy in order to maintain oxygen saturation (SpO2) greater than 94 percent (%) and is maintained up to Day 28.
Mortality Rate | Up to 28 days
Time to Sustained Clinical Improvement or Discharge From Hospital | Up to 28 days
  Sustained clinical improvement is defined as a 2-point improvement on the 8-point ordinal scale for clinical improvement, that is at least 2 points increase from the lowest score recorded since randomization and no worsening of the score afterwards by Day 28. An 8-point ordinal scale for clinical improvement in COVID-19 symptoms ranges from a score of 1 to a score of 8, where 1 (death), 2 (hospitalized, on invasive mechanical ventilation or ECMO), 3 (hospitalized, on non-invasive ventilation or high-flow oxygen devices), 4 (hospitalized, requiring supplemental oxygen), 5 (hospitalized, not requiring supplemental oxygen, requiring ongoing medical care [COVID-19 related or otherwise]), 6 (hospitalized, not requiring supplemental oxygen, no longer requires ongoing medical care), 7 (not hospitalized, limitation on activities and/or requiring home oxygen), and 8 (not hospitalized, no limitations on activities).
Time to Sustained Clinical Recovery | Up to 28 days
  Sustained clinical recovery is defined as achieving score 6, 7, or 8 based on the ordinal scale and maintained the clinical recovery until Day 28. An 8-point ordinal scale for clinical improvement in COVID-19 symptoms ranges from a score of 1 to a score of 8, where 1 (death), 2 (hospitalized, on invasive mechanical ventilation or ECMO), 3 (hospitalized, on non-invasive ventilation or high-flow oxygen devices), 4 (hospitalized, requiring supplemental oxygen), 5 (hospitalized, not requiring supplemental oxygen, requiring ongoing medical care [COVID-19 related or otherwise]), 6 (hospitalized, not requiring supplemental oxygen, no longer requires ongoing medical care), 7 (not hospitalized, limitation on activities and/or requiring home oxygen), and 8 (not hospitalized, no limitations on activities).
Percentage of Participants With Any Form of New Ventilation Use | Up to 28 days
Number of Days of New Ventilation Use | Up to 28 days
Number of Ventilation-free Days | Up to 28 days
Number of Days Free of Invasive Mechanical Ventilation or Extracorporeal Membrane Oxygenation (ECMO) | Up to 28 days
Time to Sustained Remission of Respiratory Symptoms | Up to 28 days
  Remission of respiratory symptoms is defined as independence from supplemental oxygen therapy in order to maintain SpO2 greater than 94%.
Percentage of Participants Admitted to Intensive Care Unit (ICU) | Up to 28 days
Number of Days of ICU Stay | Up to 28 days
Change From Baseline in Sequential Organ Failure Assessment (SOFA) Score at Days 7, 14, and 28 | Baseline, Days 7, 14, and 28
  The SOFA score is a scale for describing multiple organ failure in the critical care setting. It is calculated using the functional status of several organ systems: respiratory, coagulation, liver, cardiovascular, central nervous system, and renal. Each of these organ systems is rated on a scale of 1 to 4, based on objective, testable criteria, chiefly laboratory values. The ratings of each of these systems (worse observed value during that 24-hour period) are then summed to create the total score. Each organ system is assigned a point value from 0 (normal) to 4 (high degree of dysfunction/failure). The minimum score is 0, the maximum score is 24, with higher scores indicating higher likelihood of worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.